CLINICAL TRIAL: NCT01192269
Title: Buccal Cheek Cells - a New Non-invasive Fatty Acid Status Marker
Brief Title: Cheek Cells - Non-invasive Fatty Acid Status Marker
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Prof. Berthold Koletzko, Dr. von Hauner Children Hospital, Ludwig-Maximilians-Universitaet Muenchen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 116-10
Record Dates: First submitted 2010-08-16; First posted 2010-09-01 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-06

CONDITIONS: Healthy
Keywords: cheek cells; phospholipids; fatty acids; docosahexaenoic acid; Buccal Cheek cells; non invasive fatty acid status marker
MeSH Terms: interventions — Docosahexaenoic Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Docosahexaenoic Acid Supplement (Experimental): DHA supplement: Experimental
  1 x 950 mg capsules per day orally, each capsule providing ~520 mg of DHA as a triglyceride. The liquid fill contains DHASCO® oil, derived from the microalgae, Schizochytrium sp., high-oleic sunflower oil, natural mixed tocopherols, ascorbyl palmitate, and rosemary extract (flavouring). The gelatin shell contains glycerin, water, and colouring (carmel, carmine, turmeric).
  Interventions: Dietary Supplement: DHA (docosahexaenoic acid)

INTERVENTIONS:
Dietary Supplement: DHA (docosahexaenoic acid) — 1 x 950 mg capsules per day orally, each capsule providing ~520 mg of DHA as a triglyceride. The liquid fill contains DHASCO® oil, derived from the microalgae, Schizochytrium sp., high-oleic sunflower oil, natural mixed tocopherols, ascorbyl palmitate, and rosemary extract (flavouring). The gelatin shell contains glycerin, water, and colouring (carmel, carmine, turmeric).

SUMMARY:
Various biological materials have been investigated to determine dietary fatty acid intakes, such as plasma, erythrocytes, and adipose tissue. The applied techniques are invasive sampling methods and may have limitations in studies involving infants or young children. In 1985 the group of McMurchie suggested buccal cheek cells as a marker for dietary fatty acid intake; however fatty acid profiling in cheek cells has not been widely used yet.

In a clinical intervention trial a new method will be tested. The study will consist of two consecutive parts: A) a correlation study will investigate the relationship between established fatty acid markers (red blood cells (RBC), plasma) and the newly proposed markers (cheek cells) before and after intervention B) an intervention study will investigate the time depended implementation and steady state of docosahexaenoic acid DHA in plasma, RBC and cheek cells.

The participants will receive 520 mg DHA daily over a period of 30 days. Blood and cheek cell samples will be collected once prior to study commencement and regularly during intervention.

The proposed study aims at verifying cheek cell analysis results as a non-invasive marker for fatty acid profiling. This will be shown by correlation analyses of fatty acids in cheek cells, erythrocytes and plasma phospholipids. Furthermore, the time kinetics of DHA incorporation into cheek cells will clarify if cheek cell fatty acids can be considered as a short or long term marker.

The new non-invasive method is expected to be extremely valuable as a non-invasive approach for studying the fatty acid profile in human, including infants and young children. Therefore, it is of great interest to validate the new method in a clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy males and females
* Body Mass Index 20-23 kg/m2
* Average athletic activity

Exclusion Criteria:

* Fatty fish consumption > 1 per week (salmon, mackerel, sardines, herring)
* Intake of fish oil 3 months prior to study commencement
* Weight reduction diet 4 weeks prior to commencement or during intervention
* Recent (3 months prior to study commencement) medication assumed to interfere with lipid metabolism. The only exception will be the birth control pill, if the same drug (active ingredient) is taken for 3 months prior to study commencement and during the course of the study.
* Abuse of alcohol or drugs
* Pregnancy

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2010-08; Primary Completion 2011-02 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Phospholipids in buccal cheek cells | assessed basally (before intervention start) and on days 1, 2, 3, 4, 9, 14, 18, 24, 29 after the start of the intervention
  the fatty acid composition of buccal cell phospholipids and individual phospholipid species will be assessed and percentages contribution of individual fatty acids or phospholipid species, respectively, will be reported

SECONDARY OUTCOMES:
Phospholipids in plasma | assessed basally (before intervention start) and on days 1, 2, 3, 4, 9, 14, 18, 24, 29 after start of intervention
  the fatty acid composition of buccal cell phospholipids and individual phospholipid species will be assessed and percentages contribution of individual fatty acids or phospholipid species, respectively, will be reported
Phospholipids in erythrocytes | assessed basally (before intervention start) and on days 1, 2, 3, 4, 9, 14, 18, 24, 29 after start of intervention
  the fatty acid composition of buccal cell phospholipids and individual phospholipid species will be assessed and percentages contribution of individual fatty acids or phospholipid species, respectively, will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Berthold V Koletzko, MD, PhD, Principal Investigator — Dr. von Hauner Children Hospital, Ludwig-Maximilians-Universitaet Muenchen
Locations (1):
- Ludwig Maximilians University, Munich, Germany